CLINICAL TRIAL: NCT01836016
Title: Comparison of Conventional Medicine, TCM Treatment and Combination of Both Conventional Medicine and TCM Treatment for Patients With Chronic Obstructive Pulmonary Disease: A Randomized Comparative Effectiveness Research Trial
Brief Title: A Randomized Comparative Effectiveness Research Trial of Three Treatments for COPD Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER in COPD
Record Dates: First submitted 2013-04-01; First posted 2013-04-19 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Comparative effectiveness research; Medicine, Chinese Traditional; Humans; Treatment Outcome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Formoterol Fumarate; Salmeterol Xinafoate; Fluticasone; Fluticasone-Salmeterol Drug Combination; Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- conventional medicine (Experimental): According to the individualized assessment of symptoms and exacerbation risk recommended by revised 2011 GOLD, patients in this group will be given conventional medicine treatment including three drugs, which are Salbutamol (Ventolin®), Formoterol (Oxis Turbuhaler®), Salmeterol / fluticasone (Seretide®).
  Interventions: Drug: Salbutamol (Ventolin®); Drug: Formoterol (Oxis Turbuhaler®); Drug: Salmeterol / fluticasone (Seretide®)
- traditional Chinese medicine (Experimental): Patients in this group will receive four types of TCM treatment according to traditional Chinese syndrome differentiation and treatment, which are Bufei granule, Bufeijianpi granule, Bufeiyishen granule and Yiqizishen granule.
  Interventions: Drug: Bufei granule; Drug: Bufeijianpi granule; Drug: Bufeiyishen granule; Drug: Yiqizishen granule
- conventional medicine + TCM (Experimental): Patients in this group will receive conventional medicine and traditional Chinese medicine.
  Interventions: Drug: conventional medicine + TCM

INTERVENTIONS:
Drug: Salbutamol (Ventolin®) — According to the revised 2011 GOLD, patients will be divided into Group A, B, C, and D based on individualized assessment. Salbutamol was used to Group A patients for 26 weeks: Salbutamol (Ventolin®, GlaxoSmithKline) 100μg/dose, 200 inhalations. 100 μg each time (when needed), and the maximum dose is 8-12 inhalations a day.
  Other Names: Group A patients: Salbutamol (Ventolin®).
  Arms: conventional medicine
Drug: Formoterol (Oxis Turbuhaler®) — According to the revised 2011 GOLD, patients will be divided into Group A, B, C, and D based on individualized assessment. Formoterol was used to Group B patients for 26 weeks: Formoterol (Oxis Turbuhaler®, AstraZeneca), 4.5μg/ dose, 60 inhalations. 4.5μg each time, twice daily.
  Other Names: Group B patients: Formoterol (Oxis Turbuhaler®).
  Arms: conventional medicine
Drug: Salmeterol / fluticasone (Seretide®) — According to the revised 2011 GOLD, patients will be divided into Group A, B, C, and D based on individualized assessment. Salmeterol / fluticasone was used to Group C patients and Group D patients for 26 weeks: Salmeterol / fluticasone (Seretide®, GlaxoSmithKline), 50/500 μg / dose, 60 inhalations. 50/500 μg each time, twice daily.
  Other Names: Group C patients: Salmeterol / fluticasone (Seretide®).; Group D patients: Salmeterol / fluticasone (Seretide®).
  Arms: conventional medicine
Drug: Bufei granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of lung-qi deficiency will be given Bufei granule, twice daily for 26 weeks for lower dosage.
  Arms: traditional Chinese medicine
Drug: Bufeijianpi granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of deficiency of pulmonic-splenic qi will be given Bufeijianpi granule, twice daily for 26 weeks for lower dosage.
  Arms: traditional Chinese medicine
Drug: Bufeiyishen granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi of the lung and kidney will be given Bufeiyishen granule, twice daily for 26 weeks for lower dosage.
  Arms: traditional Chinese medicine
Drug: Yiqizishen granule — According to traditional Chinese syndrome differentiation and treatment, patients with syndrome of insufficiency of qi and yin of the lung and kidney will be given Yiqizishen granule, twice daily for 26 weeks for lower dosage.
  Arms: traditional Chinese medicine
Drug: conventional medicine + TCM — Patients will be given the combination of conventional medicine (Salbutamol, Formoterol, Salmeterol / fluticasone, Salmeterol / fluticasone) and (Bufei granule, Bufeijianpi granule, Bufeiyishen granule and Yiqizishen granule) for 26 weeks.
  Other Names: Both conventional medicine and traditional Chinese medicine
  Arms: conventional medicine + TCM

SUMMARY:
The aim of this study is to compare the effectiveness and economic evaluation of three treatments for Chronic Obstructive Pulmonary Disease (COPD) patients: one, conventional medicine based on 2011 Global Initiative for Chronic Obstructive Lung Disease (GOLD) and Chinese Treatment Guidelines; another, TCM treatments, which have been evaluated and have certain effect; and finally, combination of both conventional medicine and TCM treatment, then determine which treatment is the most suitable for COPD patients.

DETAILED DESCRIPTION:
COPD affects millions worldwide. The high prevalence, morbidity, mortality and economic burdens of COPD are increasing steadily. Although many therapies exist and are being developed to relieve symptoms and reduce mortality in COPD, most have only been studied in placebo-controlled efficacy studies in highly selected populations. There are few clinical trials to compare therapeutic alternatives in real world. Much of the comparative research evidence in COPD has been based on observational studies. Furthermore, studies in real world populations of COPD that received different therapies that do have efficacy evidence was found wide variations in care delivery. These considerations highlight the need to identify the most effective therapies in real world COPD patients and to design and test efforts to translate this evidence into healthcare for the millions of COPD patients. In short, there is a need for comparative effectiveness research (CER) in COPD.

CER has received growing attention worldwide. The direct comparisons of treatment alternatives provided by CER can help patients and providers make best informed treatment decisions where such evidence was previously lacking. Some randomized controlled trials on comprehensive Traditional Chinese medicine (TCM) interventions, especially based on the TCM patterns, have been the certain evidence for showing definite effect for stable COPD patients. When facing many treatment approaches, how to choose the most suitable treatment is difficult to identify. Hence, the aim of this study is to compare the effectiveness and economic evaluation of three treatments for COPD patients and then determine which treatment is the most suitable for COPD patients. conventional medicine, TCM treatment and Combination of both conventional medicine and TCM treatment.

This is a multi-center, pragmatic, randomized, controlled trial to evaluate the effectiveness of three treatments in COPD subjects. Following a 14 day run-in period, approximately 360 subjects will be randomly assigned to one of the three treatments (conventional medicine, Traditional Chinese medicine, and combination of both conventional medicine and TCM treatment) for 26 weeks. After the 26 weeks treatment period, subjects in three treatments arms will follow-up 26 weeks. The primary outcome measure is the frequency of exacerbations. and. Secondary efficacy measures include FEV1, Dyspnea (MMRC), Exercise Capacity( 6MWD), Quality of life (CAT) and economic evaluation(CEA, CUA). Safety will be assessed through the collection of adverse events. There will be a total of 5 study visits (baseline, the 13, 26 weeks of the treatment, 13 and 26 weeks of follow-up). A follow-up contact for collection of effect and economic evaluation will be conducted approximately 26 weeks following the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of mild to very severe COPD.
* medically stable
* Age between 18 and 80 years.
* Syndrome differentiation belongs to Syndrome of lung-qi deficiency, Syndrome of deficiency of pulmonic-splenic qi, Syndrome of insufficiency of qi of the lung and kidney, syndrome of insufficiency of qi and yin of the lung and kidney.
* Without participations in other interventional trials in the previous one month.
* With the informed consent signed.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study .
* Malignancy for which patient has undergone resection, radiation therapy or chemotherapy within the last 5 years.
* Current respiratory disorders other than COPD (e.g., bronchiectasis, tuberculosis, lung fibrosis, pulmonary thromboembolic).
* Complicated with heart failure (NYHA Class III or IV),or myocardial infarction within six months ,or unstable hemodynamics.
* Complicated with serious hepatic and renal diseases (liver cirrhosis, portal hypertension, bleeding of varicose veins, dialysis, or renal transplantation).
* Participating in other trials or allergic to the used medicine.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
the frequency of exacerbation | Change from Baseline in the frequency of exacerbation at Week 13 and 26 of the treatment phase, Week 13 and 26 of the follow-up phase.

SECONDARY OUTCOMES:
Forced expiratory volume in one second | Change from Baseline in FEV1 at Week 26 of the treatment phase, Week 26 of the follow-up phase.
  Forced expiratory volume in one second(FEV1) is the amount of air that can be exhaled in one second. A positive change from baseline in FEV1 indicates improvement in lung function.
Dyspnea | Change from Baseline in MMRC at Week 13 and 26 of the treatment phase, Week 13 and 26 of the follow-up phase.
  Using Modified Medical Research Council (MMRC) scale to assess a patient's level of dyspnea. The MMRC scale is a simple grading system that scored from 0 (less severe) to 4 (severe).
6 Minutes Walking Distance Test(6MWD) | Change from Baseline in 6MWD at Week 13 and 26 of the treatment phase, Week 13 and 26 of the follow-up phase.
Quality of life | Change from Baseline in CAT at Week 13 and 26 of the treatment phase, Week 13 and 26 of the follow-up phase.
  Using COPD Assessment Test ( CAT) to asses the impact of COPD on a person's life, and how this changes over time.
Economic Evaluation | 52 weeks
  Using Cost-Effective Analysis(CEA) and Cost Utility Analysis(CUA) to calculate the incremental cost-effectiveness ratio and incremental mean cost per quality-adjusted life year associated with three treatments

CONTACTS AND LOCATIONS:
Overall Officials: Jiansheng Li, MD, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Li JS, Xie Y, Li SY, Yu XQ. Comparison of conventional medicine, TCM treatment, and combination of both conventional medicine and TCM treatment for patients with chronic obstructive pulmonary disease: study protocol of a randomized comparative effectiveness research trial. Trials. 2014 May 1;15:153. doi: 10.1186/1745-6215-15-153. PMID 24885672